CLINICAL TRIAL: NCT02775240
Title: A Phase 1, Open-label, 2-period Fixed-sequence Study to Evaluate the Effect of Multiple Doses of SHP620 (Maribavir) on the Pharmacokinetics of Digoxin and Dextromethorphan in Healthy Adult Subjects
Brief Title: Study of SHP620 (Maribavir) in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SHP620-115
Record Dates: First submitted 2016-04-20; First posted 2016-05-17 (Estimated); Results first posted 2019-01-16 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Cytomegalovirus (CMV)
Keywords: Maribavir
MeSH Terms: interventions — Digoxin; maribavir; Dextromethorphan

ARMS (3):
- Digoxin (Active Comparator): On Day 1, subjects will receive a single 0.5 mg (2 x 0.25 mg) oral dose of digoxin.
  Interventions: Drug: Digoxin
- Maribavir (Experimental): On Day 8 through Day 15, subjects will receive a 400 mg (2 x 200 mg) BID oral dose of maribavir. Subjects will be given the second dose of maribavir approximately 12 hours after the first dose. On Day 13, subjects will receive a coadministration of a single 0.5 mg (2 x 0.25 mg) oral dose of digoxin and a single 30 mg oral dose of dextromethorphan given with the morning dose of maribavir.
  Interventions: Drug: Digoxin; Drug: Maribavir; Drug: Dextromethorphan
- Dextromethorphan (Active Comparator): On Day 1, subjects will receive a single 30 mg oral dose of dextromethorphan.
  Interventions: Drug: Dextromethorphan

INTERVENTIONS:
Drug: Digoxin — 0.5 mg (2 x 0.25 mg) Digoxin oral dose
  Arms: Digoxin; Maribavir
Drug: Maribavir — 200mg twice a day for 8 days
  Arms: Maribavir
Drug: Dextromethorphan — 30 mg oral dose
  Arms: Dextromethorphan; Maribavir

SUMMARY:
The purpose of this study is to determine how an investigational treatment (maribavir) is handled by the body when administered with two already approved drugs (digoxin and dextromethorphan). The study will also look at the safety and tolerability when maribavir is coadministered with digoxin and dextromethorphan versus digoxin and dextromethorphan alone.

ELIGIBILITY:
Inclusion Criteria:

* An understanding, ability, and willingness to fully comply with study procedures and restrictions.
* Ability to provide written, personally signed, and dated informed consent to participate in the study, before completing any study-related procedures.
* Age 18-50 years, inclusive at the time of consent.
* Subjects must be willing to consent to and provide blood samples for pharmacogenomics analysis.
* Willingness to comply with any applicable contraceptive requirements of the protocol and is:

  1. Male, or
  2. Female of non-childbearing potential
  3. Non-pregnant, non-lactating female
  4. Females must be at least 90 days postpartum or nulliparous.
* Must be considered "healthy." Healthy status is defined by absence of evidence of any active or chronic disease following a detailed medical and surgical history, a complete physical examination including vital signs, 12-lead ECG, hematology, blood chemistry (includes T3, T4, and TSH at screening only), and urinalysis.
* Body mass index (BMI) between 18.5 and 30.0 kg/m2 inclusive.
* Hemoglobin is equal to or greater than 12.0g/dL.
* Ability to swallow a dose of investigational product (which may be multiple tablets at one time or consecutively 1 tablet at a time)

Exclusion Criteria:

* Subject has a clinically significant history or a disorder detected during the medical interview/physical examination such as any cardiovascular, broncho-pulmonary, gastrointestinal (eg, inflammatory bowel disease, chronic diarrhea), hepatic, biliary (including gallbladder removal), renal, hematological, endocrine, autoimmune, neurological, or psychiatric disease (including depression) or any other medical condition that is capable of altering the absorption, metabolism, or elimination of drugs; or of constituting a risk factor when taking the investigational product in the judgment of the investigator.
* Known or suspected intolerance or hypersensitivity to the investigational product(s), closely related compounds, or any of the stated ingredients.
* Significant illness, as judged by the investigator, within 2 weeks of the first dose of investigational product.
* Known history of alcohol or other substance abuse within the last year.
* Donation of blood or blood products (eg, plasma or platelets) within 60 days prior to receiving the first dose of investigational product.
* Within 30 days prior to the first dose of investigational product:

  1. Have used an investigational product (if elimination half-life is <6 days, otherwise 5 half-lives).
  2. Have been enrolled in a clinical study (including vaccine studies) that, in the investigator's opinion, may impact this study.
  3. Have had any substantial changes in eating habits, as assessed by the investigator.
* Confirmed systolic blood pressure >139 mmHg or <89 mmHg and diastolic blood pressure >89 mmHg or <49 mmHg.
* Twelve-lead ECG demonstrating QTcB >450 msec at screening.
* A positive screen for alcohol or drugs of abuse at screening or Day -1, Period 1.
* Male subjects who consume more than 21 units of alcohol per week or 3 units per day; female subjects who consume more than 14 units of alcohol per week or 2 units per day (1 alcohol unit=1 beer or 1 wine [5 oz/150 mL] or 1 liquor [1.5 oz/40 mL] or 0.75 oz alcohol).
* A positive human immunodeficiency virus, hepatitis B surface antibody, or hepatitis C virus antibody screen.
* Use of tobacco in any form (eg, smoking or chewing) or other nicotine-containing products in any form (eg, gum, patch). Ex-users must report that they have stopped using tobacco for at least 30 days prior to receiving the first dose of investigational product.
* Routine consumption of more than 2 units of caffeine per day or subjects who experience caffeine withdrawal headaches. (One caffeine unit is contained in the following items: one 6 oz [180 mL] cup of coffee, two 12 oz [360 mL] cans of cola, one 12 oz cup of tea, or three 1 oz [85 g] chocolate bars. Decaffeinated coffee, tea, or cola are not considered to contain caffeine.)
* Prior screen failure, randomization, participation, or enrollment in this study or prior enrollment in a clinical study investigating maribavir.
* Current use (defined as use within 14 days prior to the first dose of investigational product) of any medication (including over-the-counter, herbal, or homeopathic preparations [eg, St. John's wort, ginkgo biloba]) with the exception of hormonal replacement therapy and occasional use of ibuprofen and acetaminophen.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Ingestion of known CYP3A modulators within 7 days of Day 1, Period 1 (includes grapefruit or grapefruit juice, oranges, Seville oranges, apples or apple juice, vegetables from the mustard green family [eg, kale, broccoli, watercress, collard greens, kohlrabi, Brussels sprouts, mustard], charbroiled meats, and products containing these ingredients).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2016-07-21 (Actual); Primary Completion 2016-09-12 (Actual); Study Completion 2016-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Clinical Pharmacology of Miami, Inc., Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Song IH, Ilic K, Murphy J, Lasseter K, Martin P. Effects of Maribavir on P-Glycoprotein and CYP2D6 in Healthy Volunteers. J Clin Pharmacol. 2020 Jan;60(1):96-106. doi: 10.1002/jcph.1504. Epub 2019 Aug 6. PMID 31385617

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in a single center in the United States between 16 August 2016 (first participant first visit) and 31 August 2016 (last participant last visit).
Pre-assignment Details: A total of 18 participants were screened and were enrolled in the study and received the treatment.
Groups:
- Treatment A and B: On Day 1, participants received a single 0.5 mg (2 × 0.25 mg) oral dose of digoxin and a single 30 mg (2 x 15 mg) oral dose of dextromethorphan (Treatment A) followed by a wash out period of minimum 7 days until start of treatment B, during which participants received maribavir 400 mg (2 x 200 mg) orally twice daily from Day 8 to Day 15. On Day 13, participants received a single 0.5 mg (2 × 0.25 mg) oral dose of digoxin and a single 30 mg (2 × 15 mg) oral dose of dextromethorphan co-administered with the morning dose of maribavir. The test product, maribavir and the investigational products, digoxin and dextromethorphan, were provided in the form of tablet.
Period: Overall Study
Arm/Group | Treatment A and B
Started | 18
Started Treatment A | 18
Started Treatment B | 17
Completed | 17
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: Safety set consisted of all participants who were administered at least 1 dose of investigational product (maribavir, digoxin, or dextromethorphan) and had at least 1 post-dose safety assessment.
Arm/Group | Treatment A and B
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: Year] | 38.1 (8.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 11

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Digoxin
Description: Cmax is the maximum observed plasma concentration of digoxin.
Time Frame: Pre-dose,0.25,0.5,1,1.5,2,3,4,5,6,8,12,24,48,72 hours post-dose on Day 1 for Treatment A and Day 13 for Treatment B
Population: Pharmacokinetic (PK) set consisted of all participants who received at least 1 dose of investigational product and had evaluable PK data (defined as complete concentration-time profile to obtain meaningful estimates of PK parameters) available for 1 dose regimen.
Measure: Geometric Mean (95% Confidence Interval); unit: Nanogram per milliliter (ng/mL)
Groups:
- Treatment A: Participants received a single 0.5 mg (2 x 0.25 mg) oral dose of digoxin tablet and a single 30 mg (2 x 15 mg) oral dose of dextromethorphan tablet on Day 1.
- Treatment B: Participants received maribavir 400 mg (2 x 200 mg) tablet orally twice daily from Day 8 to Day 15. On Day 13, participants received a single 0.5 mg (2 × 0.25 mg) oral dose of digoxin tablet and a single 30 mg (2 × 15 mg) oral dose of dextromethorphan tablet co-administered with the morning dose of maribavir.
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 18 | 17
Nanogram per milliliter (ng/mL) | 1.94 [1.60 to 2.36] | 2.35 [1.98 to 2.80]
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Comparison of Treatment B over Treatment A for Cmax of Digoxin; Test type: Other; Linear mixed effects model; Ratio of geometric means = 1.248, 90% CI 2-sided [1.130 to 1.378] — Log-transformed Cmax values were compared between treatment regimens using a linear mixed effects model with treatment regimen as fixed effect and participant as random effect

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Dextromethorphan
Description: Cmax is the maximum observed plasma concentration of dextromethorphan.
Time Frame: Pre-dose,0.25,0.5,1,1.5,2,3,4,5,6,8,12,24,48,72 hours post-dose on Day 1 for Treatment A and Day 13 for Treatment B
Population: PK set consisted of all participants who received at least 1 dose of investigational product and had evaluable PK data (defined as complete concentration-time profile to obtain meaningful estimates of PK parameters) available for 1 dose regimen.
Measure: Geometric Mean (95% Confidence Interval); unit: Nanogram per milliliter (ng/mL)
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 18 | 17
Nanogram per milliliter (ng/mL) | 1.14 [0.63 to 2.06] | 1.14 [0.65 to 1.99]
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Comparison of Treatment B over Treatment A for Cmax of Dextromethorphan; Test type: Other; Linear mixed effects model; Ratio of geometric means = 0.944, 90% CI 2-sided [0.778 to 1.144]

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Dextrorphan
Description: Cmax is the maximum observed plasma concentration of dextrorphan, the metabolite of dextromethorphan.
Time Frame: Pre-dose,0.25,0.5,1,1.5,2,3,4,5,6,8,12,24,48,72 hours post-dose on Day 1 for Treatment A and Day 13 for Treatment B
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Nanogram per milliliter (ng/mL)
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 18 | 17
Nanogram per milliliter (ng/mL) | 433 [347 to 539] | 401 [324 to 496]
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Comparison of Treatment B over Treatment A for Cmax of Dextrorphan; Test type: Other; Linear mixed effects model; Ratio of geometric means = 0.943, 90% CI 2-sided [0.883 to 1.007] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Maribavir
Description: Cmax is the maximum observed plasma concentration of maribavir.
Time Frame: Pre-dose, 0.25,0.5,1,1.5,2,3,4,5,6,8,12 hours post-dose on Day 13
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Microgram per milliliter (mcg/mL)
Arm/Group | Treatment B
Number analyzed (Participants) | 17
Microgram per milliliter (mcg/mL) | 17.6 [15.5 to 19.9]

5. Primary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Digoxin
Description: Tmax is the time to reach the maximum observed drug concentration in plasma during a dosing interval.
Time Frame: Pre-dose,0.25,0.5,1,1.5,2,3,4,5,6,8,12,24,48,72 hours post-dose on Day 1 for Treatment A and Day 13 for Treatment B
Population: as for outcome 2
Measure: Median (Full Range); unit: Hour (h)
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 18 | 17
Hour (h) | 1.00 [0.500 to 1.50] | 1.00 [0.500 to 2.00]

6. Primary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Dextromethorphan
Description: Tmax is the time to reach the maximum observed drug concentration in plasma during a dosing interval.
Time Frame: Pre-dose,0.25,0.5,1,1.5,2,3,4,5,6,8,12,24,48,72 hours post-dose on Day 1 for Treatment A and Day 13 for Treatment B
Population: as for outcome 2
Measure: Median (Full Range); unit: Hour (h)
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 18 | 17
Hour (h) | 3.00 [1.50 to 5.00] | 3.00 [2.00 to 5.00]

7. Primary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Dextrorphan
Description: Tmax is the time to reach the maximum observed drug concentration in plasma during a dosing interval.
Time Frame: Pre-dose,0.25,0.5,1,1.5,2,3,4,5,6,8,12,24,48,72 hours post-dose on Day 1 for Treatment A and Day 13 for Treatment B
Population: as for outcome 2
Measure: Median (Full Range); unit: Hour (h)
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 18 | 17
Hour (h) | 2.00 [1.50 to 3.00] | 2.00 [1.00 to 4.00]

8. Primary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Maribavir
Description: Tmax is the time to reach the maximum observed drug concentration in plasma during a dosing interval.
Time Frame: Pre-dose, 0.25,0.5,1,1.5,2,3,4,5,6,8,12 hours post-dose on Day 13
Population: as for outcome 2
Measure: Median (Full Range); unit: Hour (h)
Arm/Group | Treatment B
Number analyzed (Participants) | 17
Hour (h) | 2.00 [0.500 to 3.00]

9. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve Extrapolated to Infinity (AUC0-infinity) of Digoxin
Description: AUC0-infinity is the area under the plasma concentration versus time curve extrapolated to infinity, calculated using the observed value of the last non-zero concentration.
Time Frame: Pre-dose,0.25,0.5,1,1.5,2,3,4,5,6,8,12,24,48,72 hours post-dose on Day 1 for Treatment A and Day 13 for Treatment B
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Nanogram*hour per milliliter (ng*h/mL)
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 18 | 17
Nanogram*hour per milliliter (ng*h/mL) | 31.6 [26.9 to 37.2] | 37.3 [32.9 to 42.2]
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Comparison of Treatment B over Treatment A for AUC0-infinity of Digoxin; Test type: Other; Linear mixed effects model; Ratio of geometric means = 1.206, 90% CI 2-sided [1.099 to 1.324] — Log-transformed AUC0-infinity values were compared between treatment regimens using a linear mixed effects model with treatment regimen as fixed effect and participant as random effect

10. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve Extrapolated to Infinity (AUC0-infinity) of Dextromethorphan
Description: as for outcome 9
Time Frame: Pre-dose,0.25,0.5,1,1.5,2,3,4,5,6,8,12,24,48,72 hours post-dose on Day 1 for Treatment A and Day 13 for Treatment B
Population: as for outcome 2
Measure: Number; unit: Nanogram*hour per milliliter (ng*h/mL)
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 5 | 5
Nanogram*hour per milliliter (ng*h/mL)
  Participant 1 | 290.74 | 179.19
  Participant 2 | 28.10 | NA — Terminal phase was not available for this participant.
  Participant 3 | NA — Terminal phase was not available for this profile. | 25.14
  Participant 4 | 168.69 | 95.95
  Participant 5 | 48.33 | 41.65
  Participant 6 | 26.79 | 18.08

11. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve Extrapolated to Infinity (AUC0-infinity) of Dextrorphan
Description: as for outcome 9
Time Frame: Pre-dose,0.25,0.5,1,1.5,2,3,4,5,6,8,12,24,48,72 hours post-dose on Day 1 for Treatment A and Day 13 for Treatment B
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Nanogram*hour per milliliter (ng*h/mL)
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 18 | 17
Nanogram*hour per milliliter (ng*h/mL) | 2270 [2050 to 2520] | 2150 [1940 to 2390]
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Comparison of Treatment B over Treatment A for AUC0-infinity of Dextrorphan; Test type: Other; Linear mixed effects model; Ratio of geometric means = 0.971, 90% CI 2-sided [0.943 to 0.999] — [estimate comment as in outcome 9, analysis 1]

12. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From the Time of Dosing to the Last Measurable Concentration (AUClast) of Digoxin
Description: AUClast is the area under the plasma concentration versus time curve from the time of dosing to the last measurable concentration.
Time Frame: Pre-dose,0.25,0.5,1,1.5,2,3,4,5,6,8,12,24,48,72 hours post-dose on Day 1 for Treatment A and Day 13 for Treatment B
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Nanogram*hour per milliliter (ng*h/mL)
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 18 | 17
Nanogram*hour per milliliter (ng*h/mL) | 23.0 [19.9 to 26.6] | 26.7 [24.3 to 29.4]
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Comparison of Treatment B over Treatment A for AUClast for Digoxin; Test type: Other; Linear mixed effects model; Ratio of geometric means = 1.179, 90% CI 2-sided [1.080 to 1.287] — Log-transformed AUClast values were compared between treatment regimens using a linear mixed effects model with treatment regimen as fixed effect and participant as random effect

13. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From the Time of Dosing to the Last Measurable Concentration (AUClast) of Dextromethorphan
Description: as for outcome 12
Time Frame: Pre-dose,0.25,0.5,1,1.5,2,3,4,5,6,8,12,24,48,72 hours post-dose on Day 1 for Treatment A and Day 13 for Treatment B
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Nanogram*hour per milliliter (ng*h/mL)
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 18 | 17
Nanogram*hour per milliliter (ng*h/mL) | 7.06 [3.09 to 16.1] | 6.77 [3.02 to 15.2]
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Comparison of Treatment B over Treatment A for AUClast of Dextromethorphan; Test type: Other; Linear mixed effects model; Ratio of geometric means = 0.882, 90% CI 2-sided [0.696 to 1.118] — [estimate comment as in outcome 12, analysis 1]

14. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From the Time of Dosing to the Last Measurable Concentration (AUClast) of Dextrorphan
Description: as for outcome 12
Time Frame: Pre-dose,0.25,0.5,1,1.5,2,3,4,5,6,8,12,24,48,72 hours post-dose on Day 1 for Treatment A and Day 13 for Treatment B
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Nanogram*hour per milliliter (ng*h/mL)
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 18 | 17
Nanogram*hour per milliliter (ng*h/mL) | 2200 [1980 to 2450] | 2110 [1890 to 2360]
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Comparison of Treatment B over Treatment A for AUClast for Dextrorphan; Test type: Other; Linear mixed effects model; Ratio of geometric means = 0.973, 90% CI 2-sided [0.949 to 0.998] — [estimate comment as in outcome 12, analysis 1]

15. Primary Outcome: Parent/Metabolite Ratio of Area Under the Plasma Concentration Versus Time Curve From the Time of Dosing to the Last Measurable Concentration (AUClast) for Dextromethorphan Over AUClast for Dextrorphan (AUClast Parent/Metabolite Ratio)
Description: AUClast parent/metabolite ratio is the ratio of AUClast for dextromethorphan over AUClast for dextrorphan.
Time Frame: Pre-dose,0.25,0.5,1,1.5,2,3,4,5,6,8,12,24,48,72 hours post-dose on Day 1 for Treatment A and Day 13 for Treatment B
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio of AUClast
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 18 | 17
Ratio of AUClast | 0.003 [0.001 to 0.008] | 0.003 [0.001 to 0.008]
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Comparison of Treatment B over Treatment A for Dextromethorphan/Dextrorphan (Parent/Metabolite) AUClast ratio; Test type: Other; Linear mixed effects model; Ratio of geometric means = 0.905, 90% CI 2-sided [0.721 to 1.138] — Log-transformed AUClast ratio values were compared between treatment regimens using a linear mixed effects model with treatment regimen as fixed effect and participant as random effect

16. Primary Outcome: Parent/Metabolite Ratio of Area Under the Plasma Concentration Versus Time Curve Extrapolated to Infinity (AUC0-infinity) for Dextromethorphan Over AUC0-infinity for Dextrorphan (AUC0-infinity Parent/Metabolite Ratio)
Description: AUC0-infinity parent/metabolite ratio is the ratio of AUC0-infinity for dextromethorphan over AUC0-infinity for dextrorphan.
Time Frame: Pre-dose,0.25,0.5,1,1.5,2,3,4,5,6,8,12,24,48,72 hours post-dose on Day 1 for Treatment A and Day 13 for Treatment B
Population: as for outcome 2
Measure: Number; unit: Ratio of AUC0-infinity
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 5 | 5
Ratio of AUC0-infinity
  Participant 1 | 0.177 | 0.127
  Participant 2 | 0.009 | NA — Terminal phase was not available for this participant.
  Participant 3 | NA — Terminal phase was not available for this participant. | 0.014
  Participant 4 | 0.096 | 0.056
  Participant 5 | 0.028 | 0.025
  Participant 6 | 0.013 | 0.008

17. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time Zero to the End of the Dosing Interval at Steady-State (AUCtau) of Maribavir
Description: AUCtau is the area under the plasma concentration versus time curve from the time zero to the end of the dosing interval at steady-state.
Time Frame: Pre-dose, 0.25,0.5,1,1.5,2,3,4,5,6,8,12 hours post-dose on Day 13
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Microgram*hour per milliliter (mcg*h/mL)
Arm/Group | Treatment B
Number analyzed (Participants) | 17
Microgram*hour per milliliter (mcg*h/mL) | 91.5 [79.7 to 105]

18. Primary Outcome: First-order Rate Constant (Lambda z) Associated With the Terminal (Log-linear) Portion of the Curve of Digoxin
Description: Lambda z is the first-order rate constant associated with the terminal (log-linear) portion of the plasma concentration versus time curve, determined as the negative slope of the terminal log-linear phase of the curve.
Time Frame: Pre-dose,0.25,0.5,1,1.5,2,3,4,5,6,8,12,24,48,72 hours post-dose on Day 1 for Treatment A and Day 13 for Treatment B
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Per hour (/h)
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 18 | 17
Per hour (/h) | 0.02 [0.02 to 0.02] | 0.02 [0.01 to 0.02]

19. Primary Outcome: First-order Rate Constant (Lambda z) Associated With the Terminal (Log-linear) Portion of the Curve of Dextromethorphan
Description: as for outcome 18
Time Frame: Pre-dose,0.25,0.5,1,1.5,2,3,4,5,6,8,12,24,48,72 hours post-dose on Day 1 for Treatment A and Day 13 for Treatment B
Population: as for outcome 2
Measure: Number; unit: Per hour (/h)
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 5 | 5
Per hour (/h)
  Participant 1 | 0.04 | 0.04
  Participant 2 | 0.08 | NA — Terminal phase was not available for this participant.
  Participant 3 | NA — Terminal phase was not available for this participant. | 0.11
  Participant 4 | 0.07 | 0.08
  Participant 5 | 0.10 | 0.12
  Participant 6 | 0.10 | 0.10

20. Primary Outcome: First-order Rate Constant (Lambda z) Associated With the Terminal (Log-linear) Portion of the Curve of Dextrorphan
Description: as for outcome 18
Time Frame: Pre-dose,0.25,0.5,1,1.5,2,3,4,5,6,8,12,24,48,72 hours post-dose on Day 1 for Treatment A and Day 13 for Treatment B
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Per hour (/h)
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 18 | 17
Per hour (/h) | 0.16 [0.13 to 0.19] | 0.17 [0.14 to 0.20]

21. Primary Outcome: Terminal Half-life (t1/2) of Digoxin
Description: Terminal half-life (t1/2) is the time in hours required for the concentration of the drug to reach half of its original value.
Time Frame: Pre-dose,0.25,0.5,1,1.5,2,3,4,5,6,8,12,24,48,72 hours post-dose on Day 1 for Treatment A and Day 13 for Treatment B
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Hour (h)
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 18 | 17
Hour (h) | 41.5 [38.8 to 44.4] | 41.8 [36.7 to 47.6]

22. Primary Outcome: Terminal Half-life (t1/2) of Dextromethorphan
Description: as for outcome 21
Time Frame: Pre-dose,0.25,0.5,1,1.5,2,3,4,5,6,8,12,24,48,72 hours post-dose on Day 1 for Treatment A and Day 13 for Treatment B
Population: as for outcome 2
Measure: Number; unit: Hour (h)
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 5 | 5
Hour (h)
  Participant 1 | 15.86 | 16.17
  Participant 2 | 9.09 | NA — Terminal phase was not available for this participant.
  Participant 3 | NA — Terminal phase was not available for this participant. | 6.43
  Participant 4 | 9.82 | 8.72
  Participant 5 | 6.86 | 5.58
  Participant 6 | 6.71 | 7.03

23. Primary Outcome: Terminal Half-life (t1/2) of Dextrorphan
Description: as for outcome 21
Time Frame: Pre-dose,0.25,0.5,1,1.5,2,3,4,5,6,8,12,24,48,72 hours post-dose on Day 1 for Treatment A and Day 13 for Treatment B
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Hour (h)
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 18 | 17
Hour (h) | 4.42 [3.63 to 5.37] | 4.16 [3.55 to 4.87]

24. Primary Outcome: Terminal Half-life (t1/2) of Maribavir
Description: as for outcome 21
Time Frame: Pre-dose, 0.25,0.5,1,1.5,2,3,4,5,6,8,12 hours post-dose on Day 13
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Hour (h)
Arm/Group | Treatment B
Number analyzed (Participants) | 17
Hour (h) | 4.04 [3.66 to 4.46]

25. Primary Outcome: Apparent Oral Clearance (CL/F) of Digoxin
Description: CL/F is equal to dose/AUC0-infinity (dose divided by area under the plasma concentration versus time curve extrapolated to infinity [AUC0-infinity]).
Time Frame: Pre-dose,0.25,0.5,1,1.5,2,3,4,5,6,8,12,24,48,72 hours post-dose on Day 1 for Treatment A and Day 13 for Treatment B
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Liter per hour (L/h)
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 18 | 17
Liter per hour (L/h) | 15.8 [13.4 to 18.6] | 13.4 [11.9 to 15.2]

26. Primary Outcome: Apparent Oral Clearance (CL/F) of Dextromethorphan
Description: as for outcome 25
Time Frame: Pre-dose,0.25,0.5,1,1.5,2,3,4,5,6,8,12,24,48,72 hours post-dose on Day 1 for Treatment A and Day 13 for Treatment B
Population: as for outcome 2
Measure: Number; unit: Liter per hour (L/h)
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 5 | 5
Liter per hour (L/h)
  Participant 1 | 103.19 | 167.42
  Participant 2 | 1067.64 | NA — Terminal phase was not available for this participant.
  Participant 3 | NA — Terminal phase was not available for this participant. | 1193.51
  Participant 4 | 177.84 | 312.65
  Participant 5 | 620.71 | 720.23
  Participant 6 | 1119.90 | 1659.07

27. Primary Outcome: Apparent Oral Clearance (CL/F) of Maribavir
Description: CL/F is equal to dose/AUCtau (dose divided by area under the curve from time 0 to the end of the dosing interval at steady state [AUCtau])
Time Frame: Pre-dose, 0.25,0.5,1,1.5,2,3,4,5,6,8,12 hours post-dose on Day 13
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Liter per hour (L/h)
Arm/Group | Treatment B
Number analyzed (Participants) | 17
Liter per hour (L/h) | 2.19 [1.90 to 2.51]

28. Primary Outcome: Concentration at the End of Dosing Interval (Ctau) of Maribavir
Description: Ctau is the concentration of maribavir at the end of the dosing interval.
Time Frame: Pre-dose, 0.25,0.5,1,1.5,2,3,4,5,6,8,12 hours post-dose on Day 13
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Microgram per milliliter (mcg/mL)
Arm/Group | Treatment B
Number analyzed (Participants) | 17
Microgram per milliliter (mcg/mL) | 2.13 [1.66 to 2.73]

29. Primary Outcome: Volume of Distribution Divided by the Fraction of Dose Absorbed (Vz/F) of Digoxin
Description: Vz/F is the volume of distribution associated with the terminal slope following extravascular administration divided by the fraction of dose absorbed.
Time Frame: Pre-dose,0.25,0.5,1,1.5,2,3,4,5,6,8,12,24,48,72 hours post-dose on Day 1 for Treatment A and Day 13 for Treatment B
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Liter (L)
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 18 | 17
Liter (L) | 946 [804 to 1110] | 809 [723 to 906]

30. Primary Outcome: Volume of Distribution Divided by the Fraction of Dose Absorbed (Vz/F) of Dextromethorphan
Description: as for outcome 29
Time Frame: Pre-dose,0.25,0.5,1,1.5,2,3,4,5,6,8,12,24,48,72 hours post-dose on Day 1 for Treatment A and Day 13 for Treatment B
Population: as for outcome 2
Measure: Number; unit: Liter (L)
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 5 | 5
Liter (L)
  Participant 1 | 2360.54 | 3904.44
  Participant 2 | 14008.68 | NA — Terminal phase was not available for this participant.
  Participant 3 | NA — Terminal phase was not available for this participant. | 11078.42
  Participant 4 | 2519.11 | 3931.63
  Participant 5 | 6142.85 | 5796.87
  Participant 6 | 10836.77 | 16835.78

31. Primary Outcome: Pre-dose Concentration (C0) of Maribavir
Description: C0 is the lowest concentration reached by a drug before the next dose is administered.
Time Frame: Pre-dose on Day 13
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Microgram per milliliter (mcg/mL)
Arm/Group | Treatment B
Number analyzed (Participants) | 17
Microgram per milliliter (mcg/mL) | 2.64 [1.92 to 3.62]

32. Secondary Outcome: Number of Participants With Study-related Adverse Events (AEs), Serious Adverse Events (SAEs) and Treatment-emergent Adverse Events (TEAEs)
Description: An AE was any untoward medical occurrence in a participant administered an investigational product (IP) and that did not necessarily have a causal relationship with this treatment. AE was considered to be study-related if there was any valid reason, even if undetermined or untested, for suspecting a possible cause-and-effect relationship between the IP and the occurrence of the AE. An AE was considered a TEAE if it had a start date on or after the first dose of IP or if it had a start date before the date of the first dose of IP, but increased in intensity on or after the date of the first dose of IP. A serious adverse event (SAE) was any untoward medical occurrence (related either to the test product or to the other IP or not) that at any dose resulted in death; was life-threatening; required or prolongation of hospitalization; resulted in persistent or significant disability/incapacity; was a congenital abnormality/birth defect; was an important medical event.
Time Frame: From start of study drug administration up to follow-up (up to 25 days)
Population: Safety set consisted of all participants who were administered at least 1 dose of the test product (maribavir) or to the other investigational products (digoxin and dextrometorphan) and had at least 1 post-dose safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 18 | 17
Participants
  Study related TEAE | 4 | 12
  Serious AE | 0 | 0
  Any TEAE | 4 | 12

33. Secondary Outcome: Number of Participants With Clinically Significant Changes Reported as TEAE in Physical Examination, Vital Signs, 12-lead ECGs, Hematology, Blood Chemistry and Urinalysis
Description: Clinical significance of the changes observed in the safety parameters to be reported as TEAE was interpreted by the investigator.
Time Frame: Baseline up to Day 16
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 18 | 17
Participants
  Physical examination | 0 | 0
  Vital signs | 0 | 0
  12-lead ECGs | 0 | 0
  Hematology | 0 | 0
  Blood Chemistry | 0 | 0
  Urinalysis | 0 | 0

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to follow-up (up to 25 days)
Arm/Group | Treatment A | Treatment B
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/17
Other Adverse Events (participants affected / at risk) | 4/18 | 12/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A (N=18) | Treatment B (N=17)
Dry eye (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 7 (8)
Headache (Nervous system disorders) | 2 (2) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.